CLINICAL TRIAL: NCT03525093
Title: A Hypnotherapeutic Group Training to Improve Coping With Perceived Stress - a Prospective Controlled Interventional Multicenter Trial
Brief Title: Hypnotherapy to Improve Coping With Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Benno Brinkhaus, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYPNOSTRESS2
Record Dates: First submitted 2018-04-23; First posted 2018-05-15 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis + health education (Active Comparator): 5 sessions of group hypnosis, each 90 minutes; plus CDs/MP3 recordings to train at home plus health education booklet on coping with stress
  Interventions: Behavioral: Hypnosis
- Health education alone (Other): Patients receive a health education booklet to improve coping with stress
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Hypnosis — 5 session of group hypnosis, each 90 minutes, to reduce subjective levels of stress, improve coping with stress. Additional audiotapes of hypnosis sessions as homework.
  Participants receive a health education booklet on improving coping with stress.
  Arms: Hypnosis + health education
Behavioral: Health education — Participants receive a health education booklet on improving coping with stress.
  Arms: Health education alone

SUMMARY:
This prospective controlled study aims to test a 5 week group hypnosis training as intervention to improve coping with perceived psychological stress.

ELIGIBILITY:
Inclusion Criteria:

* Healthy or health-stable participants between 18 and 65 years with increased perceived stress for at least 3 months
* Perceived stress in the last week on the visual analog scale> 40 mm (VAS 0 - 100 mm)
* Ability to consent and sign declaration of consent

Exclusion Criteria:

* Current or planned participation in a stress management exercise within the next 17 weeks
* Current use of psychotherapeutic treatment
* Presence of moderate or severe acute or chronic disease
* Presence of an acute or chronic mental disorder
* Participation in a study within the last 2 months prior to enrollment
* Lack of understanding of the German language

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Perceived Stress on Visual Analogue Scale | 5 weeks
  Visual Analogue Scale of perceived stress in the last week, 0-100 mm (0=no stress; 100 = extreme stress)

SECONDARY OUTCOMES:
Perceived Stress on Visual Analogue Scale | 12 weeks
  Visual Analogue Scale of perceived stress in the last week, 0-100 mm (0=no stress; 100 = extreme stress)
Cohens Perceived Stress Scale 10 Items | 5 weeks, 12 weeks
  Cohen S, Kamarck T, and Mermelstein R, "A global measure of perceived stress," Journal of Health and Social Behavior, vol. 24, no. 4, pp. 385-396, 1983.
Stress reduction on Likert Scale | 5 weeks, 12 weeks
  Stress rating on a Likert Scale
Allgemeine Depressionsskala (ADS-K) | 5 weeks, 12 weeks
  Hautzinger M, Bailer M, Hofmeister D, Keller F. (2012). Allgemeine Depressionsskala (ADS) (2. Aufl.). Göttingen: Hogrefe.
General Self Efficacy Scale (Schwarzer) | 5 weeks, 12 weeks
  Schwarzer R, Jerusalem M. (Hrsg.). Skalen zur Erfassung von Lehrer- und Schülermerkmalen: Dokumentation der psychometrischen Verfahren im Rahmen der Wissenschaftlichen Begleitung des Modellversuchs Selbstwirksame Schulen. Berlin: Freie Universität Berlin, 1999.
SF 36 Quality of Life | 5 weeks, 12 weeks
  Bullinger M, Kirchberger I: SF-36: Fragebogen zum Gesundheitszustand, Hogrefe, Göttingen, Germany, 1998.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité University Berlin, Berlin, Germany

REFERENCES:
- [Derived] Siewert J, Teut M, Brinkhaus B, Fisch S, Kummer S. The relevance of outcome expectations in group hypnosis for stress reduction: a secondary analysis of a multicenter randomized controlled trial. Front Psychol. 2024 Apr 19;15:1363037. doi: 10.3389/fpsyg.2024.1363037. eCollection 2024. PMID 38708017
- [Derived] Fisch S, Trivakovic-Thiel S, Roll S, Keller T, Binting S, Cree M, Brinkhaus B, Teut M. Group hypnosis for stress reduction and improved stress coping: a multicenter randomized controlled trial. BMC Complement Med Ther. 2020 Nov 13;20(1):344. doi: 10.1186/s12906-020-03129-6. PMID 33187503